CLINICAL TRIAL: NCT05518604
Title: Pregnancy, Active Duty and Weight Loss (PADaWL) Study: A Randomized Controlled Trial Assessing the Effect of Dietary Intervention on Postpartum Weight Loss in Active Duty Women
Brief Title: Weight Loss and Physical Fitness Following Pregnancy in Active Duty Women
Acronym: PADaWL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Gehrich MD, Obstetrician and Gynecologist, Urogynecologist, Minimally Invasive Gynecologic Surgeon, Tripler Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-15411
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Weight Loss; Postpartum Weight Retention
Keywords: Weight loss; Exercise; Diet; Physical Fitness; Postpartum; Active Duty
MeSH Terms: conditions — Weight Loss; Gestational Weight Gain; Motor Activity | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Active Duty women will be enrolled during pregnancy and randomized postpartum to one of three groups for the first year postpartum.
  Group 1- dietary counseling with close monitoring utilizing a biometric fitness device Group 2- Close monitoring with biometric fitness device Group 3 Routine postpartum care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Arm 1 (Experimental): Women in this arm will undergone dietary counseling in the first year postpartum in addition to close supervision of diet, exercise, and sleep.
  Interventions: Behavioral: Counseling with goal of modifying eating behaviors
- Intervention Arm 2 (Experimental): Women in this arm will not have dietary counseling but will have close supervision of diet, exercise and sleep.
  Interventions: Behavioral: Counseling with goal of modifying eating behaviors
- Control (No Intervention): Women in this arm will undergo routine postpartum care.

INTERVENTIONS:
Behavioral: Counseling with goal of modifying eating behaviors — Dietary counseling will occur virtually a minimum of 4x and as desired by participant in the first year postpartum according to a standard protocol
  Arms: Intervention Arm 1; Intervention Arm 2

SUMMARY:
Pregnancy and delivery are major stressors on the female body and contribute significantly to permanent weight gain and associated morbidity in women. This can profoundly affect the ability of active duty (AD) women to advance in their career. The first 12 weeks postpartum are the time period during which the most significant weight loss occurs and is critical in achieving a healthy weight in the first year postpartum. Many factors contribute to effective weight loss in this period among which the most critical are diet, exercise, and sleep. Breast feeding and depression may also affect weight changes postpartum. Research has shown diet to likely be the most crucial of these factors.

The PADaWL study is designed as a randomized controlled trial to assess the effects of dietary intervention on weight and physical fitness versus routine postpartum care in the first year postpartum. Subjects will be primiparous AD women from any military service recruited in the obstetric clinic in the third trimester of pregnancy at Tripler Army Medical Center. Data will collected in an ambi-directional fashion with pre-pregnancy physical fitness data, demographic and pregnancy data collected at time of enrollment. Subjects will be randomized to receive intensive virtual sessions with a dietician vs routine postpartum care for the first 12 months postpartum. We will utilize a biometric device to monitor activity levels and sleep, web-based diaries to monitor breast feeding and diet, and validated questionnaires to evaluate depression as well as diet and sleep. Subjects will be monitored weekly for the first 12 weeks postpartum and will then be further evaluated at 6, 9 and 12 months postpartum.

Primary outcome is weight at 12weeks postpartum and whether subjects have achieved military standards. Secondary outcome will be weight at 12 months postpartum and whether subject has achieved weight and fitness standards. The study intends to collect large amounts of data, and we intend to analyze which factors may be contributing to weight retention postpartum.

This study should provide an accurate assessment of the effects of pregnancy on AD women. It should generate a clean and accurate dataset on which multiple follow-on studies can be performed and provide data for designing further intervention studies in postpartum women. The results of this study should also be able to assist in developing policy and guidance concerning AD women and pregnancy.

DETAILED DESCRIPTION:
RESEARCH BACKGROUND:

Women naturally gain weight beyond that of the added pregnancy tissue and many gradually lose this excess weight following delivery. In the US, 15-27% of women across all ethnic groups have excess postpartum weight retention (PPWR) of > 10lbs one year after delivery. (Lipsky, Strawderman, and Olson 2012, 1496-1502); (Gunderson et al. 2008, 178-187); (DeGroot et al. 2021a, e0255248) This issue has also been documented in AD women across multiple services with 12-15% not meeting fitness standards at one year postpartum. (DeGroot et al. 2021b, e0255248) (Rogers et al. 2020, e227-e234) This is an immediate concern for AD women as it has a detrimental effect on career progression. Weight retention also has long-term consequences for health including contributing significantly to the risk of obesity, diabetes, heart disease and hypertension. It is shown that women who return to their pre-pregnancy weight by about six months have a lower risk of being overweight 10 years later. (Amorim Adegboye and Linne 2013, CD005627) This critical postpartum time period in a woman's life has major repercussions on her well-being. A significant number of women are never able to effectively lose weight and achieve fitness postpartum. Long-term, the added weight and resulting metabolic effects of postpartum weight retention lead to chronic health conditions such as obesity type II diabetes, chronic hypertension and other components of metabolic syndrome. (Linne et al. 2003, 1516-1522) Many AD women succumb to this cycle of weight retention and are unable to serve effectively in the military. This affects 10-20% of AD women who become pregnant while serving and was highlighted by retrospective research performed at Tripler Army Medical Center. (DeGroot et al. 2021a, e0255248) Our literature review reveals five factors that contribute significantly to weight changes following delivery in AD women: diet, exercise, breastfeeding, sleep and depression.

RESEARCH GOALS AND OBJECTIVES:

The PADaWL study seeks to determine if dietary interventions by a licensed dietician in the first year postpartum will lead to more effective weight loss and ultimately physical fitness than routine postpartum care among a cohort of AD service members.

The primary goal of this research is to determine how effectively AD women lose weight and recover fitness after delivery. Specifically, aims of this study are to:

Aim#1: Identify factors that influence the timing of active duty servicewomen return-to-duty fitness postpartum.

Aim #2: Characterize the utility of a biometric device to monitor multi-factorial influences on achieving pre-pregnancy fitness postpartum Aim #3: Determine the effectiveness of intensive dietary counseling in the first year postpartum on weight loss and physical fitness.

STUDY PROCEDURES:

I. Recruitment will be performed using multiple methods and can be recruited at any time during their pregnancy: Passive recruitment will occur in the TAMC OB/GYN clinic. Posters will be displayed throughout the OB/GYN clinic with tabs showing phone numbers allowing the patients to contact researchers directly to inquire about the study. Active recruitment will occur in the TAMC OB/GYN clinic. Providers will directly ask AD women who are obstetric patients whether they are interested in participating and direct them to the research staff. If necessary, appointments in MHS Genesis will be screened for healthy primiparous AD women with an uncomplicated singleton pregnancy who would be candidates for the study.

II. Screening for Eligibility: Potential participants will be approached and screened for inclusion and exclusion criteria by either one of the researchers or research assistants. This will be done via telephone call. If they are interested in participating in the study, they will be sent a flyer detailing the study via email. If they maintain interest in participating in the study, they will be asked to meet with the research team at the time of their 34-37week appointment.

III. Enrollment: Eligible potential participants will meet a member of the research team either before or after their 34-37week appointment. They will bring a copy of their pre- pregnancy fitness report. During this appointment they will be rescreened. Informed Consent and HIPPA consent will be obtained. Randomization will occur. Subjects will be assigned a de-identified study subject number. An anonymous myfitnesspal.com account will be opened, and they will be asked to familiarize themselves with the website. Subjects will be asked to obtain a scale for home use. Subject will be given a hand- out on all the data which will be collected on her during the course of the study.

IV. Data collection at Enrollment: After signing the consent, subjects will be asked to complete questionnaires on fitness and diet during their pregnancy. These questionnaires will be on-line, and they will enter their data utilizing their anonymous study ID. A demographic, cultural and social questionnaire will be obtained.

V. Retrospective Data collected after Enrollment: Weight gain in pregnancy, Conditions complicating pregnancy, EPDS score at 28weeks VI. Delivery: All AD women participants in the PADaWL study coming to TAMC L&D for their delivery after 35 weeks will be identified based on the posted website list, via screening of patients on the postpartum ward, or will contact research personnel via telephone call or text. Lipid profile labs will be drawn at the time of their admission with the remainder of their obstetric labs. Subjects will deliver their newborn and after stabilization will be transferred to the postpartum ward. On postpartum day #1 or #2, the subject will be approached by the research team in the postpartum ward. Subjects will be given the Garmin fitness tracker and given instructions on use. The subject will use their initials and only their birthday year to set up the app. She will be asked to start recording diet and activity levels (primarily measured as steps and caloric expenditure) on the day after being discharged from hospital. She will be given repeat instructions on appropriate monitoring of diet and exercise. Before discharge she will obtain a 6-week postpartum appointment with one the researchers. Intervention group will obtain their first virtual nutrition counseling appointment to occur within the first month postpartum VII. Randomized groups to active vs routine dietary management: Both groups will receive the following: Nutrition education handouts pertaining to healthy postpartum eating, Nutrition education handouts pertaining to calorie counting procedures to include websites, apps, and methods of estimating caloric intake, General calorie recommendations based on participant age, height, weight, and activity level Intervention group will receive: One-on-one appointments with a Registered Dietitian via virtual health within the first month postpartum, three months postpartum, six months postpartum, and 12 months postpartum VIII. First 12 weeks postpartum: Period of intense data collection: All subjects will be collecting daily diet information via myfitnesspal.com. All subjects will be collecting activity as well as sleep levels via the Garmin fitness tracker. This data will be downloaded automatically to the website via their smart phone. All subjects will document her breast feeding weekly in the myfitnesspal.com app. All subjects will obtain weekly weights and place data onto their myfitnesspal.com website. The intervention group will have a virtual nutrition counseling appointment within the first month postpartum and a second appointment in the third month postpartum. At the 6- week postpartum appointment with one of the research investigators, subjects will submit a EPDS questionnaire to assess depression. This weekly data will be collected through their 12weeks postpartum. The data will be accessible by the research personnel via the internet. If data is missing, the subject will be contacted by research personnel to improve compliance.

IX. 6 months postpartum: Subjects will undergo telephonic interview with research team. The following data will be obtained: Weight, Dietary questionnaire, Fitness questionnaire, Sleep questionnaire, EPDS, Breast feeding data, The intervention group will have a 3rd virtual nutrition counseling in this timeframe.

X. 9 months postpartum: The intervention group will undergo a fourth and final virtual nutrition counseling appointment in this timeframe.

XI. 12 months postpartum: The patient will undergo her first military fitness evaluation for record at 1 year postpartum including weight and height. She will be asked to bring a copy of these data to her 12month postpartum visit.

XII. 12 months postpartum: Subjects will undergo a clinic visit with physical exam with one of the research investigators. In addition, they will submit the following data: Weight, Dietary questionnaire, Fitness questionnaire, Sleep questionnaire, EPDS, Breast feeding data, Post-study questionnaire. The intervention group will have a final virtual nutrition counseling appointment.

STAISTICAL ANALYSIS

Aim#1:

The outcomes evaluated are 1) the ability of AD women to achieve military weight standards at 12 weeks, 6months and 1 year postpartum, and 2) improvement in mandated physical fitness assessment at 12 months postpartum.

Odds ratio and t-test will be used to compare pre-pregnancy and postpartum fitness results for the collective enrollment. ANOVA with repeated measures over time will be used to evaluate differences between pre pregnancy, at delivery, and different time points post pregnancy for weight. Regression analysis will be used to determine the linear regression algorithm for weight loss over time for each participant from delivery through up to one year postpartum to determine the x intercept of the time point when weight equals pre pregnancy weight for each participant. This time period of return to pre pregnancy weight can be used along with percent weight loss at 12 weeks post pregnancy as the metrics to examine the relationship with other variables of sleep, breast feeding, activity, etc.Multiple variate stepwise regression analysis will be used to identify which variables most strongly independently influence weight loss (period of time before pre pregnancy weight is achieved, and/or percent weight loss at specific timepoints (1eg. 2 weeks, 6 months, 1 year) from delivery date). Which variables are covariates with other variables will also be determined.

Aim #2:

The efficacy of the fitness tracker to monitor postpartum women as they regain fitness in the year after pregnancy will be evaluated based on 1) the ability to generate consistent useable data, and 2) the acceptance by the study participants as a wearable device Descriptive statistics will be used to characterize how many events of interrupted data or non-collected data missing data occurs each week for 12 weeks postpartum Aim #3: Determine the effectiveness of intensive dietary counseling in the first year postpartum on weight loss and physical fitness.

To test the effectiveness of dietary intervention the participants will be randomized to two groups. Group 1 (n=32) will receive routine postpartum care. Group 2 (n=32) will receive dietary interventions by a licensed dietician. The metric for efficacy of the intervention will be detecting an effect size of 20% in weight, sleep score, breast feeding score ANOVA will be used to compare the two groups with repeated measures over time at 16 time points over time (pre-pregnancy, time of delivery, weekly for 12 weeks, 6 months and 12 months postpartum) for weight, sleep score, breast feeding score. For fitness and activity ANOVA at two time points (pre-pregnancy and 12 months postpartum) by group interaction effect will be analyzed.

An addendum was approved on 27 AUG 2025 in which we ask participants in the PADaWL study to undergo physiologic testing at the Armed Forces Wellness Center at between 12-18 weeks postpartum and 1 year postpartum. These phyisologic tests will be measuring body fat % and CO2 max. These data will be included in the analysis. This part of the protocol is optional for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Active Duty from any service - Army, Navy, Air Force, Marine, Coast Guard.
2. Any rank
3. Singleton Pregnancy
4. Delivery between 36weeks and 41weeks EGA
5. Non obese (<30BMI) at NOB appointment in 1st trimester.
6. Any type of delivery (spontaneous vaginal delivery, operative vaginal delivery, cesarean delivery)
7. First term pregnancy
8. Live birth
9. Must have documented standardized fitness evaluation for record prior to pregnancy
10. Must have plan to remain on AD for a minimum of 18 months following delivery.
11. Not planning short interval pregnancy within 18 months of delivery
12. Must be planning on staying on Oahu for a minimum of 12 months following delivery

Exclusion Criteria:

1. Obese ( > 30 BMI) at NOB appointment in 1st trimester
2. Delivery before 36 weeks
3. Severe maternal morbidity requiring prolonged ( > 1week) postpartum admission
4. NICU admission > 2 week
5. Profile beyond pregnancy profile limiting ability to exercise or take physical fitness exam.
6. Desires to take a leave of duty or separation from duty in the first 18 months following pregnancy
7. No physical fitness test for record in the year prior to pregnancy.
8. Prior pregnancy beyond 20 weeks
9. Planning future pregnancy within 18 months of delivery

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be female
Enrollment: 74 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Return to required weight for active duty women at 12 weeks postpartum | 12 weeks
  Primary outcome is the number of active duty women who are able to return to required weight at 12 weeks following delivery
Return to physical fitness at 12 months postpartum as assessed by physical fitness testing. | 12 months
  Secondary outcome is the number of active duty women who pass their physical fitness assessment at 1 year postpartum. This assessment includes weight and physical fitness

CONTACTS AND LOCATIONS:
Overall Officials: Alan P Gehrich, MD, Principal Investigator — Tripler Army Medical Center
Locations (2):
- United States (2):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Desmond Doss Health Clinic, Schofield Barracks, Hawaii

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amorim Adegboye AR, Linne YM. Diet or exercise, or both, for weight reduction in women after childbirth. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD005627. doi: 10.1002/14651858.CD005627.pub3. PMID 23881656
- [Background] Armitage NH, Severtsen BM, Vandermause R, Smart DA. Training for the Air Force fitness assessment: the experience of postpartum women. Mil Med. 2014 Jul;179(7):766-72. doi: 10.7205/MILMED-D-13-00437. PMID 25003862
- [Background] Armitage NH, Smart DA. Changes in Air Force fitness measurements pre- and post-childbirth. Mil Med. 2012 Dec;177(12):1519-23. doi: 10.7205/milmed-d-12-00248. PMID 23397699
- [Background] Bazzazian S, Riazi H, Vafa M, Mahmoodi Z, Nasiri M, Mokhtaryan-Gilani T, Ozgoli G. The relationship between depression, stress, anxiety, and postpartum weight retention: A systematic review. J Educ Health Promot. 2021 Jun 30;10:230. doi: 10.4103/jehp.jehp_1409_20. eCollection 2021. PMID 34395667
- [Background] Berger AA, Peragallo-Urrutia R, Nicholson WK. Systematic review of the effect of individual and combined nutrition and exercise interventions on weight, adiposity and metabolic outcomes after delivery: evidence for developing behavioral guidelines for post-partum weight control. BMC Pregnancy Childbirth. 2014 Sep 10;14:319. doi: 10.1186/1471-2393-14-319. PMID 25208549
- [Background] Bijlholt M, Van Uytsel H, Ameye L, Devlieger R, Bogaerts A. Eating behaviors in relation to gestational weight gain and postpartum weight retention: A systematic review. Obes Rev. 2020 Oct;21(10):e13047. doi: 10.1111/obr.13047. Epub 2020 Jun 1. PMID 32476253
- [Background] Blaine BE, Rodman J, Newman JM. Weight loss treatment and psychological well-being: a review and meta-analysis. J Health Psychol. 2007 Jan;12(1):66-82. doi: 10.1177/1359105307071741. PMID 17158841
- [Background] Blau LE, Hormes JM. Preventing Excess Gestational Weight Gain and Obesity in Pregnancy: the Potential of Targeting Psychological Mechanisms. Curr Obes Rep. 2020 Dec;9(4):522-529. doi: 10.1007/s13679-020-00415-9. Epub 2020 Nov 4. PMID 33145706
- [Background] Chauhan SP, Johnson TL, Magann EF, Woods JY, Chen HY, Sheldon IV, Morrison JC. Compliance with regulations on weight gain 6 months after delivery in active duty military women. Mil Med. 2013 Apr;178(4):406-11. doi: 10.7205/MILMED-D-12-00394. PMID 23707825
- [Background] Dalrymple KV, Flynn AC, Relph SA, O'Keeffe M, Poston L. Lifestyle Interventions in Overweight and Obese Pregnant or Postpartum Women for Postpartum Weight Management: A Systematic Review of the Literature. Nutrients. 2018 Nov 7;10(11):1704. doi: 10.3390/nu10111704. PMID 30405088
- [Background] DeGroot DW, Sitler CA, Lustik MB, Langan KL, Hauret KG, Gotschall MH, Gehrich AP. The effect of pregnancy and the duration of postpartum convalescence on the physical fitness of healthy women: A cohort study of active duty servicewomen receiving 6 weeks versus 12 weeks convalescence. PLoS One. 2021 Jul 28;16(7):e0255248. doi: 10.1371/journal.pone.0255248. eCollection 2021. PMID 34320030
- [Background] Dewey KG, Lovelady CA, Nommsen-Rivers LA, McCrory MA, Lonnerdal B. A randomized study of the effects of aerobic exercise by lactating women on breast-milk volume and composition. N Engl J Med. 1994 Feb 17;330(7):449-53. doi: 10.1056/NEJM199402173300701. PMID 8289849
- [Background] Elliott-Sale KJ, Barnett CT, Sale C. Systematic review of randomised controlled trials on exercise interventions for weight management during pregnancy and up to one year postpartum among normal weight, overweight and obese women. Pregnancy Hypertens. 2014 Jul;4(3):234. doi: 10.1016/j.preghy.2014.03.015. Epub 2014 Jul 9. PMID 26104620
- [Background] Endres LK, Straub H, McKinney C, Plunkett B, Minkovitz CS, Schetter CD, Ramey S, Wang C, Hobel C, Raju T, Shalowitz MU; Community Child Health Network of the Eunice Kennedy Shriver National Institute of Child Health and Human Development. Postpartum weight retention risk factors and relationship to obesity at 1 year. Obstet Gynecol. 2015 Jan;125(1):144-152. doi: 10.1097/AOG.0000000000000565. PMID 25560116
- [Background] Goldstein RF, Abell SK, Ranasinha S, Misso M, Boyle JA, Black MH, Li N, Hu G, Corrado F, Rode L, Kim YJ, Haugen M, Song WO, Kim MH, Bogaerts A, Devlieger R, Chung JH, Teede HJ. Association of Gestational Weight Gain With Maternal and Infant Outcomes: A Systematic Review and Meta-analysis. JAMA. 2017 Jun 6;317(21):2207-2225. doi: 10.1001/jama.2017.3635. PMID 28586887
- [Background] Goldstein RF, Abell SK, Ranasinha S, Misso ML, Boyle JA, Harrison CL, Black MH, Li N, Hu G, Corrado F, Hegaard H, Kim YJ, Haugen M, Song WO, Kim MH, Bogaerts A, Devlieger R, Chung JH, Teede HJ. Gestational weight gain across continents and ethnicity: systematic review and meta-analysis of maternal and infant outcomes in more than one million women. BMC Med. 2018 Aug 31;16(1):153. doi: 10.1186/s12916-018-1128-1. PMID 30165842
- [Background] Greer JA, Zelig CM, Choi KK, Rankins NC, Chauhan SP, Magann EF. Return to military weight standards after pregnancy in active duty working women: comparison of marine corps vs. navy. J Matern Fetal Neonatal Med. 2012 Aug;25(8):1433-7. doi: 10.3109/14767058.2011.639820. Epub 2012 Apr 3. PMID 22081961
- [Background] Gunderson EP, Rifas-Shiman SL, Oken E, Rich-Edwards JW, Kleinman KP, Taveras EM, Gillman MW. Association of fewer hours of sleep at 6 months postpartum with substantial weight retention at 1 year postpartum. Am J Epidemiol. 2008 Jan 15;167(2):178-87. doi: 10.1093/aje/kwm298. Epub 2007 Oct 29. PMID 17971337
- [Background] He X, Zhu M, Hu C, Tao X, Li Y, Wang Q, Liu Y. Breast-feeding and postpartum weight retention: a systematic review and meta-analysis. Public Health Nutr. 2015 Dec;18(18):3308-16. doi: 10.1017/S1368980015000828. Epub 2015 Apr 21. PMID 25895506
- [Background] Hill B, McPhie S, Skouteris H. The Role of Parity in Gestational Weight Gain and Postpartum Weight Retention. Womens Health Issues. 2016 Jan-Feb;26(1):123-9. doi: 10.1016/j.whi.2015.09.012. Epub 2015 Nov 3. PMID 26542383
- [Background] Hill CC, Gloeb DJ. Military maternal weight trends and perinatal outcomes. Mil Med. 2013 Aug;178(8):880-6. doi: 10.7205/MILMED-D-13-00031. PMID 23929049
- [Background] Hoover EA, Louis JM. Optimizing Health: Weight, Exercise, and Nutrition in Pregnancy and Beyond. Obstet Gynecol Clin North Am. 2019 Sep;46(3):431-440. doi: 10.1016/j.ogc.2019.04.003. Epub 2019 Jun 21. PMID 31378286
- [Background] Lasikiewicz N, Myrissa K, Hoyland A, Lawton CL. Psychological benefits of weight loss following behavioural and/or dietary weight loss interventions. A systematic research review. Appetite. 2014 Jan;72:123-37. doi: 10.1016/j.appet.2013.09.017. Epub 2013 Sep 27. PMID 24075862
- [Background] Lim S, O'Reilly S, Behrens H, Skinner T, Ellis I, Dunbar JA. Effective strategies for weight loss in post-partum women: a systematic review and meta-analysis. Obes Rev. 2015 Nov;16(11):972-87. doi: 10.1111/obr.12312. Epub 2015 Aug 27. PMID 26313354
- [Background] Linne Y, Dye L, Barkeling B, Rossner S. Weight development over time in parous women--the SPAWN study--15 years follow-up. Int J Obes Relat Metab Disord. 2003 Dec;27(12):1516-22. doi: 10.1038/sj.ijo.0802441. PMID 14634683
- [Background] Linne Y, Rossner S. Interrelationships between weight development and weight retention in subsequent pregnancies: the SPAWN study. Acta Obstet Gynecol Scand. 2003 Apr;82(4):318-25. doi: 10.1080/j.1600-0412.2003.00150.x. PMID 12716315
- [Background] Lipsky LM, Strawderman MS, Olson CM. Maternal weight change between 1 and 2 years postpartum: the importance of 1 year weight retention. Obesity (Silver Spring). 2012 Jul;20(7):1496-502. doi: 10.1038/oby.2012.41. Epub 2012 Feb 15. PMID 22334257
- [Background] Makama M, Skouteris H, Moran LJ, Lim S. Reducing Postpartum Weight Retention: A Review of the Implementation Challenges of Postpartum Lifestyle Interventions. J Clin Med. 2021 Apr 27;10(9):1891. doi: 10.3390/jcm10091891. PMID 33925502
- [Background] Mannan M, Doi SA, Mamun AA. Association between weight gain during pregnancy and postpartum weight retention and obesity: a bias-adjusted meta-analysis. Nutr Rev. 2013 Jun;71(6):343-52. doi: 10.1111/nure.12034. Epub 2013 May 2. PMID 23731445
- [Background] Marangoni F, Cetin I, Verduci E, Canzone G, Giovannini M, Scollo P, Corsello G, Poli A. Maternal Diet and Nutrient Requirements in Pregnancy and Breastfeeding. An Italian Consensus Document. Nutrients. 2016 Oct 14;8(10):629. doi: 10.3390/nu8100629. PMID 27754423
- [Background] McCrory MA, Nommsen-Rivers LA, Mole PA, Lonnerdal B, Dewey KG. Randomized trial of the short-term effects of dieting compared with dieting plus aerobic exercise on lactation performance. Am J Clin Nutr. 1999 May;69(5):959-67. doi: 10.1093/ajcn/69.5.959. PMID 10232637
- [Background] McKinley MC, Allen-Walker V, McGirr C, Rooney C, Woodside JV. Weight loss after pregnancy: challenges and opportunities. Nutr Res Rev. 2018 Dec;31(2):225-238. doi: 10.1017/S0954422418000070. Epub 2018 Jul 9. PMID 29984681
- [Background] Miller MJ, Kutcher J, Adams KL. Effect of Pregnancy on Performance of a Standardized Physical Fitness Test. Mil Med. 2017 Nov;182(11):e1859-e1863. doi: 10.7205/MILMED-D-17-00093. PMID 29087853
- [Background] Nascimento SL, Pudwell J, Surita FG, Adamo KB, Smith GN. The effect of physical exercise strategies on weight loss in postpartum women: a systematic review and meta-analysis. Int J Obes (Lond). 2014 May;38(5):626-35. doi: 10.1038/ijo.2013.183. Epub 2013 Sep 19. PMID 24048142
- [Background] Pedersen P, Baker JL, Henriksen TB, Lissner L, Heitmann BL, Sorensen TI, Nohr EA. Influence of psychosocial factors on postpartum weight retention. Obesity (Silver Spring). 2011 Mar;19(3):639-46. doi: 10.1038/oby.2010.175. Epub 2010 Aug 12. PMID 20706201
- [Background] Phelan S. Pregnancy: a "teachable moment" for weight control and obesity prevention. Am J Obstet Gynecol. 2010 Feb;202(2):135.e1-8. doi: 10.1016/j.ajog.2009.06.008. Epub 2009 Aug 15. PMID 19683692
- [Background] Phelan S, Hagobian T, Brannen A, Hatley KE, Schaffner A, Munoz-Christian K, Tate DF. Effect of an Internet-Based Program on Weight Loss for Low-Income Postpartum Women: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2381-2391. doi: 10.1001/jama.2017.7119. PMID 28632867
- [Background] Rauh K, Gunther J, Kunath J, Stecher L, Hauner H. Lifestyle intervention to prevent excessive maternal weight gain: mother and infant follow-up at 12 months postpartum. BMC Pregnancy Childbirth. 2015 Oct 15;15:265. doi: 10.1186/s12884-015-0701-2. PMID 26472133
- [Background] Rogers AE, Khodr ZG, Bukowinski AT, Conlin AMS, Faix DJ, Garcia SMS. Postpartum Fitness and Body Mass Index Changes in Active Duty Navy Women. Mil Med. 2020 Feb 12;185(1-2):e227-e234. doi: 10.1093/milmed/usz168. PMID 31295347
- [Background] Ruchat SM, Mottola MF, Skow RJ, Nagpal TS, Meah VL, James M, Riske L, Sobierajski F, Kathol AJ, Marchand AA, Nuspl M, Weeks A, Gray CE, Poitras VJ, Jaramillo Garcia A, Barrowman N, Slater LG, Adamo KB, Davies GA, Barakat R, Davenport MH. Effectiveness of exercise interventions in the prevention of excessive gestational weight gain and postpartum weight retention: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1347-1356. doi: 10.1136/bjsports-2018-099399. PMID 30337461
- [Background] Ryan RA, Lappen H, Bihuniak JD. Barriers and Facilitators to Healthy Eating and Physical Activity Postpartum: A Qualitative Systematic Review. J Acad Nutr Diet. 2022 Mar;122(3):602-613.e2. doi: 10.1016/j.jand.2021.11.015. Epub 2021 Nov 25. PMID 34839027
- [Background] Siega-Riz AM, Herring AH, Carrier K, Evenson KR, Dole N, Deierlein A. Sociodemographic, perinatal, behavioral, and psychosocial predictors of weight retention at 3 and 12 months postpartum. Obesity (Silver Spring). 2010 Oct;18(10):1996-2003. doi: 10.1038/oby.2009.458. Epub 2009 Dec 24. PMID 20035283
- [Background] Stahlman S, Witkop CT, Clark LL, Taubman SB. Pregnancies and live births, active component service women, U.S. Armed Forces, 2012-2016. MSMR. 2017 Nov;24(11):2-9. PMID 29211489
- [Background] Stendell-Hollis NR, Thompson PA, West JL, Wertheim BC, Thomson CA. A comparison of Mediterranean-style and MyPyramid diets on weight loss and inflammatory biomarkers in postpartum breastfeeding women. J Womens Health (Larchmt). 2013 Jan;22(1):48-57. doi: 10.1089/jwh.2012.3707. Epub 2012 Dec 31. PMID 23276189
- [Background] van der Pligt P, Willcox J, Hesketh KD, Ball K, Wilkinson S, Crawford D, Campbell K. Systematic review of lifestyle interventions to limit postpartum weight retention: implications for future opportunities to prevent maternal overweight and obesity following childbirth. Obes Rev. 2013 Oct;14(10):792-805. doi: 10.1111/obr.12053. Epub 2013 Jun 17. PMID 23773448
- [Background] van Poppel MN, Hartman MA, Hosper K, van Eijsden M. Ethnic differences in weight retention after pregnancy: the ABCD study. Eur J Public Health. 2012 Dec;22(6):874-9. doi: 10.1093/eurpub/cks001. Epub 2012 Feb 7. PMID 22315462
- [Background] Walker LO, Sterling BS, Kim M, Arheart KL, Timmerman GM. Trajectory of weight changes in the first 6 weeks postpartum. J Obstet Gynecol Neonatal Nurs. 2006 Jul-Aug;35(4):472-81. doi: 10.1111/j.1552-6909.2006.00062.x. PMID 16881991
- [Background] Wambach K, Spencer B: Breastfeeding and human lactation. Sixth edition. ed. Burlington, MA: Jones & Bartlett Learning; 2021. Includes bibliographical references and index.; ID: alma9917448023406676.
- [Background] Weina SU. Effects of pregnancy on the Army Physical Fitness Test. Mil Med. 2006 Jun;171(6):534-7. doi: 10.7205/milmed.171.6.534. PMID 16808137
- [Background] Wilkinson SA, van der Pligt P, Gibbons KS, McIntyre HD. Trial for Reducing Weight Retention in New Mums: a randomised controlled trial evaluating a low intensity, postpartum weight management programme. J Hum Nutr Diet. 2015 Jan;28 Suppl 1:15-28. doi: 10.1111/jhn.12193. Epub 2013 Nov 25. PMID 24267102
- [Background] Xiao RS, Kroll-Desrosiers AR, Goldberg RJ, Pagoto SL, Person SD, Waring ME. The impact of sleep, stress, and depression on postpartum weight retention: a systematic review. J Psychosom Res. 2014 Nov;77(5):351-8. doi: 10.1016/j.jpsychores.2014.09.016. Epub 2014 Oct 2. PMID 25306538